CLINICAL TRIAL: NCT04333589
Title: The Mechanism, Clinical Outcome and Therapeutic Intervention of Corona Virus Disease 2019 Patients Whose Nucleic Acids Changed From Negative to Positive
Brief Title: Corona Virus Disease 2019 Patients Whose Nucleic Acids Changed From Negative to Positive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Guiqiang Wang, Principal Investigator, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020 research 112
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Favipiravir
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir group (Experimental): On the 1st day, 1600mg each time, twice a day; from the 2nd to the 7th day, 600mg each time, twice a day. Oral administration, the maximum number of days taken is not more than 14 days.
  Interventions: Drug: Favipiravir
- Regular treatment group (No Intervention): Treatments other than lopinavir and ritonavir, chloroquine phosphate, hydroxychloroquine sulfate, arbidol, and colomycin can be given.

INTERVENTIONS:
Drug: Favipiravir — On the 1st day, 1600mg each time, twice a day; from the 2nd to the 7th day, 600mg each time, twice a day. Oral administration, the maximum number of days taken is not more than 14 days.
  Arms: Favipiravir group

SUMMARY:
To investigate the mechanism, clinical outcome and therapeutic efficacy with favipiravir of Corona Virus Disease 2019 patients whose nucleic acids changed from negative to positive.

DETAILED DESCRIPTION:
In clinical institutions that enroll corona virus disease 2019 patients whose nucleic acids changed from negative to positive, two arms, multi-center, randomized and controlled methods are adopted. Patients are divided into two groups, favipiravir group and regular treatment group. 210 patients are expected to be enrolled and the cases are allocated according to the ratio of 2( favipiravir group): 1(regular treatment group).

ELIGIBILITY:
Inclusion Criteria:

1. COVID-19 has been diagnosed, and the nucleic acid test of respiratory specimens such as sputum or nasopharyngeal swabs has been negative for two consecutive times after treatment (sampling time interval of at least 24 hours);
2. The nucleic acid test of specimens such as sputum, throat swabs, blood, feces and other specimens was positive for COVID-19 during screening visits;
3. Voluntarily participate in research and sign informed consent.

Exclusion Criteria:

1. Those allergic to fapilavir;
2. Pregnant or lactating women;
3. Unstable liver, kidney, and heart diseases;
4. History of mental disorders, substance abuse or dependence;
5. Researchers consider it inappropriate to participate in research;
6. Participating in other clinical research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Viral nucleic acid test negative conversion rate | 5 months
  Proportion of subjects who tested negative for nucleic acid from sputum or nasopharyngeal swabs for two consecutive times(sampling time at least 24 hours).

SECONDARY OUTCOMES:
Clinical cure rate | 5 months
  Definition of clinical cure: The viral load of the respiratory specimen was negative for two consecutive times (the interval between the two tests was greater than or equal to one day), the lung image improved, and the body temperature returned to normal for more than 3 days, and the clinical manifestation improved.

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, Principal Investigator — Peking University First Hospital
Locations (8):
- China (8):
  - The Second People's Hospital of Fuyang, Fuyang, Anhui
  - Ezhou Hospital of Traditional Chinese Medicine, Ezhou, Hubei
  - Ezhou Central Hospital, Wuhan, Hubei
  - Huoshenshan Hospital of Wuhan, Wuhan, Hubei
  - Jinyintan Hospital of Wuhan, Wuhan, Hubei
  - Wuhan Pulmonary Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Wenzhou Medical University Affiliated First Hospital, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Li J, Zhang C, Wu Z, Wang G, Zhao H. The Mechanism and Clinical Outcome of patients with Corona Virus Disease 2019 Whose Nucleic Acid Test has changed from negative to positive, and the therapeutic efficacy of Favipiravir: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jun 5;21(1):488. doi: 10.1186/s13063-020-04430-y. PMID 32503657